CLINICAL TRIAL: NCT04828993
Title: A SINGLE ARM, MULTICENTER, OPEN-LABEL STUDY TO EVALUATE THE EFFICACY, SAFETY, TOLERABILITY, AND PHARMACODYNAMICS OF ORALLY ADMINISTERED TAFAMIDIS MEGLUMINE IN TRANSTHYRETIN AMYLOID POLYNEUROPATHY PARTICIPANTS IN CHINA
Brief Title: The Effect Of Tafamidis Meglumine In Transthyretin Amyloid Polyneuropathy Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B3461078
Record Dates: First submitted 2021-03-17; First posted 2021-04-02 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Transthyretin Amyloid Polyneuropathy (ATTR-PN)
Keywords: tafamidis meglumine
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tafamidis treatment arm (Experimental): Chinese patients diagnosed with ATTR-PN treated with tafamidis 20mg once daily oral administration for 72 weeks (18 months).
  Interventions: Drug: tafamidis meglumine

INTERVENTIONS:
Drug: tafamidis meglumine — Tafamidis meglumine 20 mg, once daily, oral administration, for 72 weeks (18 months).
  Other Names: Vyndaqel

SUMMARY:
This is a single-arm, open-label, multicenter study designed to evaluate the efficacy, safety, tolerability as well as pharmacodynamics of tafamidis meglumine in ATTR-PN participants in China.

Approximately 10-15 participants are planned to be enrolled. All enrolled participants will receive oral tafamidis meglumine 20 mg soft capsules once daily for 72 weeks (18 months).

DETAILED DESCRIPTION:
This is a single-arm, open-label, multicenter study designed to evaluate the efficacy, safety, tolerability as well as pharmacodynamics of tafamidis meglumine in ATTR-PN participants in China.

All enrolled participants will receive oral tafamidis meglumine 20 mg soft capsules once daily starting on Day 1. Clinical visits will be scheduled at Baseline (Day 1) and at Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60 and Week 72. At Week 36 and Week 60 site visit, assessment of adverse events, safety related lab testings, concomitant medications and investigational product compliance will be scheduled. Every 6 weeks (do not exceed 7 weeks since last confirmation) telephone contacts will be made during visits in which no investigative site visits are scheduled for assessment of adverse events, concomitant medications and investigational product compliance (between Week 12 and 24, between Week 24 and 36, between Week 36 and 48, between Week 48 and 60, and between Week 60 and 72).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants between the ages of 18 and 80 years.
2. Participants have amyloid documented by biopsy
3. Participants must have a TTR mutation that is associated with ATTR-PN.
4. Participants have peripheral and/or autonomic neuropathy
5. Stages of disease according to symptom severity-stage I.

Exclusion Criteria:

1. Other acute or chronic medical or psychiatric condition including recent or active suicidal ideation or behavior or laboratory abnormality, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
2. Chronic use of non-protocol approved non-steroidal anti-inflammatory drugs.
3. Use of diflunisal, tauroursodeoxycholate, doxycycline, inotersen, patisiran or any other TTR stabilizing agent, or experimental interventions for familial amyloidosis within 30 days prior to the study entry and/or during study participation. Participants who are taking or who have previously taken tafamidis.

   Prior/Concurrent Clinical Study Experience:
4. Previous administration with an investigational drug within 30 days or 5 half lives preceding the first dose of investigational product used in this study (whichever is longer).
5. Participant has primary (light chain) or secondary amyloidosis.
6. If female, participant is pregnant or breast feeding, or plans to be pregnant or breast feeding in the next 18 months.
7. Participant has received prior liver or any other organ except cornea transplantation.
8. Participant requires significant assistance with ambulation or is wheel chair bound.
9. Participants with cardiomyopathy specific TTR mutations.
10. Participant has other causes of sensorimotor neuropathy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2023-02-12 (Actual); Study Completion 2023-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- China (8):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - NanFang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Peking union hospital of Chinese academy of medical sciences, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - Tiantan Hospital Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B3461078

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 15 participants were screened and assigned to treatment.
Groups:
- Tafamidis Meglumine 20 mg Once Daily (QD): All enrolled participants received a once-daily (QD) oral dose of tafamidis meglumine 20 mg in a soft capsule formulation.
Period: Disposition Phase: TREATMENT
Arm/Group | Tafamidis Meglumine 20 mg Once Daily (QD)
Started | 15
Completed | 15
Not Completed | 0
Period: Disposition Phase: FOLLOW-UP
Arm/Group | Tafamidis Meglumine 20 mg Once Daily (QD)
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tafamidis Meglumine 20 mg Once Daily (QD)
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.1 (15.75)
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 6
  45-64 years | 5
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Neuropathy Impairment Score-lower Limb (NIS-LL) Total Score at Week 72
Description: NIS-LL: assess muscle weakness, reflexes, sensation; scored separately for left and right limbs. Components of muscle weakness (hip and knee flexion, hip and knee extension, ankle dorsiflexors, ankle plantar flexors, toe extensors, toe flexors) scored on scale 0 (normal) to 4 (paralysis), higher score=greater weakness. Components of reflexes (quadriceps femoris, triceps surae); sensation (touch pressure, pin-prick, vibration, joint position) scored 0 = normal, 1 = decreased, or 2 = absent. Total possible NIS-LL score range 0-88, high score = more impairment. Components of muscle weakness are scored to eight levels: 0 = Normal, 1 = 25% Weak, 2 = 50% Weak, 3 = 75% Weak, 3.25 = Move against gravity, 3.5 = Movement, gravity eliminated, 3.75 = Muscle flicker, no movement, 4 = Paralysis.
Time Frame: Baseline, Week 72
Population: All participants who took at least 1 dose of tafamidis meglumine soft gelatin capsule 20 mg.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Tafamidis Meglumine 20 mg Once Daily (QD)
Number analyzed (Participants) | 15
Units on a scale | 2.3 [-3.0 to 46.0]

2. Secondary Outcome: Change From Baseline in Neuropathy Impairment Score-lower Limb (NIS-LL) Total Score at Weeks 24, and 48
Description: as for outcome 1
Time Frame: Baseline, Week 24, Week 48
Population: All participants who took at least 1 dose of tafamidis meglumine soft gelatin capsule 20 mg.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Tafamidis Meglumine 20 mg Once Daily (QD)
Number analyzed (Participants) | 15
Units on a scale
  Change From Baseline in Neuropathy Impairment Score-lower limb (NIS-LL) Total Score at Week 24 | 3.0 [-20.0 to 20.0]
  Change From Baseline in Neuropathy Impairment Score-lower limb (NIS-LL) Total Score at Week 48: number analyzed (Participants) | 9
  Change From Baseline in Neuropathy Impairment Score-lower limb (NIS-LL) Total Score at Week 48 | 8.0 [-13.5 to 18.0]

3. Secondary Outcome: Change From Baseline in Total Quality of Life (TQOL) of Norfolk Quality of Life - Diabetic Neuropathy (Norfolk QOL-DN) at Weeks 24, 48, and 72
Description: Norfolk QOL-DN: 35-item participant-rated questionnaire assess the impact of neuropathy on the quality of life of participants diagnosed with transthyretin amyloid (ATTR). Scoring is based on 35 questions that yield a TQOL as well as 5 subscale scores: activities of daily living, large fiber neuropathy/physical functioning, small fiber neuropathy, autonomic neuropathy, and symptoms. TQOL= sum of all the items, total possible score range= -2 to 138, where higher score=worse quality of life.
Time Frame: Baseline, Week 24, Week 48, Week 72
Population: All participants who took at least 1 dose of tafamidis meglumine soft gelatin capsule 20 mg.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Tafamidis Meglumine 20 mg Once Daily (QD)
Number analyzed (Participants) | 15
Units on a scale
  Change From Baseline in TQOL of Norfolk QOL-DN at Week 24 | -1.00 [-26.00 to 54.00]
  Change From Baseline in TQOL of Norfolk QOL-DN at Week 48 | 2.00 [-26.00 to 63.00]
  Change From Baseline in TQOL of Norfolk QOL-DN at Week 72 | 8.00 [-11.00 to 74.00]

4. Secondary Outcome: Change From Baseline in 5 Domains of Norfolk QOL-DN at Weeks 24, 48, and 72
Description: Norfolk QOL-DN: 35-item participant-rated questionnaire assess the impact of neuropathy on the quality of life of participants diagnosed with transthyretin amyloid (ATTR). It is summarized in 5 domains: (1) Activities of daily living (score ranges from 0 to 20, where higher score=worse quality of life); (2) Large fiber neuropathy/physical functioning (score ranges from -2 to 58, where higher score=worse condition); (3) Small fiber neuropathy (score ranges from 0 to 16, where higher score=worse condition); (4) Autonomic neuropathy (score ranges from 0 to 12, where higher score=worse condition) and (5) Symptoms (score ranges from 0 to 32, where higher score=less symptoms of disease). Total possible score range= -2 to 138, where higher score=worse quality of life.
Time Frame: Baseline, Week 24, Week 48, Week 72
Population: All participants who took at least 1 dose of tafamidis meglumine soft gelatin capsule 20 mg.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Tafamidis Meglumine 20 mg Once Daily (QD)
Number analyzed (Participants) | 15
Units on a scale
  Change From Baseline in Physical Functioning/Large Fiber Domain of Norfolk QOL-DN at Week 24 | -3.00 [-22.00 to 28.00]
  Change From Baseline in Physical Functioning/Large Fiber Domain of Norfolk QOL-DN at Week 48 | 2.00 [-13.00 to 38.00]
  Change From Baseline in Physical Functioning/Large Fiber Domain of Norfolk QOL-DN at Week 72 | 4.00 [-10.00 to 39.00]
  Change From Baseline in Activities of Daily Living Domain of Norfolk QOL-DN at Week 24 | 0.00 [-4.00 to 12.00]
  Change From Baseline in Activities of Daily Living Domain of Norfolk QOL-DN at Week 48 | 1.00 [-4.00 to 15.00]
  Change From Baseline in Activities of Daily Living Domain of Norfolk QOL-DN at Week 72 | 3.00 [-2.00 to 15.00]
  Change From Baseline in Symptoms Domain of Norfolk QOL-DN at Week 24 | 1.00 [-13.00 to 9.00]
  Change From Baseline in Symptoms Domain of Norfolk QOL-DN at Week 48 | 2.00 [-6.00 to 9.00]
  Change From Baseline in Symptoms Domain of Norfolk QOL-DN at Week 72 | 2.00 [-2.00 to 23.00]
  Change From Baseline in Small Fiber Domain of Norfolk QOL-DN at Week 24 | 0.00 [-3.00 to 6.00]
  Change From Baseline in Small Fiber Domain of Norfolk QOL-DN at Week 48 | 1.00 [-2.00 to 9.00]
  Change From Baseline in Small Fiber Domain of Norfolk QOL-DN at Week 72 | 3.00 [-3.00 to 10.00]
  Change From Baseline in Autonomic Domain of Norfolk QOL-DN at Week 24 | 0.00 [-4.00 to 3.00]
  Change From Baseline in Autonomic Domain of Norfolk QOL-DN at Week 48 | 0.00 [-5.00 to 4.00]
  Change From Baseline in Autonomic Domain of Norfolk QOL-DN at Week 72 | 2.00 [-5.00 to 6.00]

5. Secondary Outcome: Change From Baseline in Modified Body Mass Index (mBMI) at Weeks 4, 8, 12, 24, 36, 48, and 72
Description: BMI is calculated by weight divided by height squared and measured as kilogram per square meter (kg/m^2). mBMI is calculated by multiplying BMI by serum albumin levels [gram/liter (g/L)]. mBMI is measured as kg/m^2*g/L. A progressive decline in mBMI indicates worsening of disease severity.
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, 48, and 72
Population: All participants who took at least 1 dose of tafamidis meglumine soft gelatin capsule 20 mg.
Measure: Median (Full Range); unit: kg/m^2*g/L
Arm/Group | Tafamidis Meglumine 20 mg Once Daily (QD)
Number analyzed (Participants) | 15
kg/m^2*g/L
  Change From Baseline in mBMI at Week 4: number analyzed (Participants) | 14
  Change From Baseline in mBMI at Week 4 | -5.9 [-87.2 to 95.5]
  Change From Baseline in Modified Body Mass Index (mBMI) at Week 8: number analyzed (Participants) | 14
  Change From Baseline in Modified Body Mass Index (mBMI) at Week 8 | 22.3 [-101.2 to 219.7]
  Change From Baseline in Modified Body Mass Index (mBMI) at Week 12 | 9.2 [-39.0 to 199.3]
  Change From Baseline in Modified Body Mass Index (mBMI) at Week 24 | 21.8 [-132.8 to 179.1]
  Change From Baseline in Modified Body Mass Index (mBMI) at Week 36: number analyzed (Participants) | 12
  Change From Baseline in Modified Body Mass Index (mBMI) at Week 36 | 37.0 [-79.3 to 207.7]
  Change From Baseline in Modified Body Mass Index (mBMI) at Week 48 | 41.4 [-130.2 to 152.6]
  Change From Baseline in Modified Body Mass Index (mBMI) at Week 72: number analyzed (Participants) | 11
  Change From Baseline in Modified Body Mass Index (mBMI) at Week 72 | 9.4 [-161.8 to 179.5]

6. Secondary Outcome: Change From Baseline in Physical Component Summary and Mental Component Summary of 36-Item Short Form Survey (SF-36) at Weeks 24, 48, and 72
Description: The SF-36 is a participant administered scale assessing general quality of life. It consists of self-administered 36-item questionnaire that measured 8 health domains: physical function, role-physical, bodily pain, general health, vitality, social function, role-emotional, and mental health. These 8 domains are also summarized as physical and mental component scores. The score for each domain and component score is the mean of the individual question scores, which are scaled from 0 (minimum) to 100 (maximum), where high scores in each dimension and high overall scores indicate a better quality of life.
Time Frame: Baseline, Weeks 24, 48, and 72
Population: All participants who took at least 1 dose of tafamidis meglumine soft gelatin capsule 20 mg.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Tafamidis Meglumine 20 mg Once Daily (QD)
Number analyzed (Participants) | 15
Units on a scale
  Change from Baseline in Physical Component Summary at Week 24: number analyzed (Participants) | 14
  Change from Baseline in Physical Component Summary at Week 24 | -2.15 [-9.29 to 11.84]
  Change from Baseline in Physical Component Summary at Week 48: number analyzed (Participants) | 14
  Change from Baseline in Physical Component Summary at Week 48 | -0.12 [-12.13 to 12.08]
  Change from Baseline in Physical Component Summary at Week 72: number analyzed (Participants) | 14
  Change from Baseline in Physical Component Summary at Week 72 | -1.60 [-17.61 to 8.89]
  Change from Baseline in Mental Component Summary at Week 24: number analyzed (Participants) | 14
  Change from Baseline in Mental Component Summary at Week 24 | 1.21 [-9.56 to 19.30]
  Change from Baseline in Mental Component Summary at Week 48: number analyzed (Participants) | 14
  Change from Baseline in Mental Component Summary at Week 48 | -2.56 [-31.69 to 9.36]
  Change from Baseline in Mental Component Summary at Week 72: number analyzed (Participants) | 14
  Change from Baseline in Mental Component Summary at Week 72 | -6.10 [-31.85 to 8.17]

7. Secondary Outcome: Change From Baseline in EuroQoL 5 Dimensions 5 Levels (EQ-5D-5L) Index Score at Weeks 24, 48, and 72
Description: EQ-5D-5L: standardized participant (aged >17 years) completed questionnaire consists of 2 components: a health state profile and an optional VAS. EQ-5D health state profile has 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems. Responses to 5 dimensions comprise a health state/a single utility index value. E.g. if a participant responds "no problems" for each 5 dimensions, then health state was coded as "11111" with a predefined index value to it. Every health state (coded as combination of responses on each of 5 dimensions) has a unique predefined utility index value assigned to it, by EuroQol. Chinese value sets (with all possible health states) is used for adults in the study, range from -0.391 to 1. Higher (positive) scores = better health state.
Time Frame: Baseline, Weeks 24, 48, and 72
Population: All participants who took at least 1 dose of tafamidis meglumine soft gelatin capsule 20 mg.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Tafamidis Meglumine 20 mg Once Daily (QD)
Number analyzed (Participants) | 15
Units on a scale
  Change from Baseline in EQ-5D-5L Index Score at Week 24 | 0.00 [-0.50 to 0.22]
  Change from Baseline in EQ-5D-5L Index Score at Week 48 | -0.05 [-0.51 to 0.11]
  Change from Baseline in EQ-5D-5L Index Score at Week 72 | -0.16 [-0.75 to 0.11]

8. Secondary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Treatment emergent adverse event is defined as any adverse event started after the first dose. The TEAEs were collected until Week 77.
Time Frame: Baseline up to Week 77
Population: All participants who took at least 1 dose of tafamidis meglumine soft gelatin capsule 20 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis Meglumine 20 mg Once Daily (QD)
Number analyzed (Participants) | 15
Participants | 13

9. Secondary Outcome: Number of Participants With Categorical Vital Signs Data
Description: Vital signs categorical criteria: 1) pulse rate <40 beats per minute (bpm), or >120 bpm; 2) standing diastolic blood pressure (BP) <50 mmHg, or increase ≥20 mmHg, or decrease ≥20 mmHg; 3) standing systolic BP <90 mmHg, or increase ≥30 mmHg, or decrease ≥30 mmHg; 4) supine diastolic BP <50 mmHg, or increase ≥20 mmHg, or decrease ≥20 mmHg; 5) supine systolic BP <90 mmHg, or increase ≥30 mmHg, or decrease ≥30 mmHg.
Time Frame: Baseline up to Week 72
Population: All participants who took at least 1 dose of tafamidis meglumine soft gelatin capsule 20 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis Meglumine 20 mg Once Daily (QD)
Number analyzed (Participants) | 15
Participants
  Pulse rate <40 bpm | 0
  Pulse rate >120 bpm | 0
  Standing diastolic BP <50 mmHg | 4
  Standing diastolic BP increase ≥20 mmHg | 3
  Standing diastolic BP decrease ≥20 mmHg | 0
  Standing systolic BP <90 mmHg | 6
  Standing systolic BP increase ≥30 mmHg | 5
  Standing systolic BP decrease ≥30 mmHg | 3
  Supine diastolic BP <50 mmHg: number analyzed (Participants) | 14
  Supine diastolic BP <50 mmHg | 0
  Supine diastolic BP increase ≥20 mmHg: number analyzed (Participants) | 14
  Supine diastolic BP increase ≥20 mmHg | 2
  Supine diastolic BP decrease ≥20 mmHg: number analyzed (Participants) | 14
  Supine diastolic BP decrease ≥20 mmHg | 2
  Supine systolic BP <90 mmHg: number analyzed (Participants) | 14
  Supine systolic BP <90 mmHg | 0
  Supine systolic BP increase ≥30 mmHg: number analyzed (Participants) | 14
  Supine systolic BP increase ≥30 mmHg | 1
  Supine systolic BP decrease ≥30 mmHg: number analyzed (Participants) | 14
  Supine systolic BP decrease ≥30 mmHg | 1

10. Secondary Outcome: Number of Participants With Categorical Electrocardiogram (ECG) Data
Description: ECG categorical criteria: 1) ECG mean heart rate <40 beats/minute, or >120 beats/minute; 2) PR interval not otherwise specified ≥300 milliseconds (msec), or baseline >200 msec and %increase ≥25%/ baseline ≤200 msec and %increase ≥50% (% change ≥25/50%); 3) QRS interval not otherwise specified ≥140 msec, or %change ≥50%; 4) QT interval not otherwise specified ≥500 msec; 5) corrected QT (QTc) interval not otherwise specified ≥450 and <480 msec, or ≥480 and <500 msec, or ≥500 msec; or change ≥30 and <60 msec, or change ≥60 msec.
Time Frame: Baseline up to Week 72
Population: All participants who took at least 1 dose of tafamidis meglumine soft gelatin capsule 20 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis Meglumine 20 mg Once Daily (QD)
Number analyzed (Participants) | 15
Participants
  ECG mean heart rate <40 beats/minute | 0
  ECG mean heart rate >120 beats/minute | 0
  PR interval not otherwise specified ≥300 milliseconds (msec) | 0
  PR interval not otherwise specified % change ≥25/50% | 0
  QRS interval not otherwise specified ≥140 msec | 1
  QRS interval not otherwise specified %change ≥50% | 1
  QT interval not otherwise specified ≥500 msec | 0
  corrected QT (QTc) interval not otherwise specified ≥450 and <480 msec | 9
  corrected QT (QTc) interval not otherwise specified ≥480 and <500 msec | 7
  corrected QT (QTc) interval not otherwise specified ≥500 msec | 3
  corrected QT (QTc) interval not otherwise specified change ≥30 and <60 msec | 5
  corrected QT (QTc) interval not otherwise specified change ≥60 msec | 1

11. Secondary Outcome: Number of Participants With Clinically Significant Echocardiography (ECHO) Value Related to Primary Diagnosis (Transthyretin Amyloidosis [ATTR]) at Baseline, Weeks 24, 48, and 72
Description: Clinically significant ECHO findings include: left ventricular (LV) posterior wall thickness greater than or equal to (>=)13 mm, LV septal thickness >= 13 mm, right ventricular thickness >= 7 mm, ratio of peak mitral early diastolic and atrial contraction velocity (E/A ratio) >= 2, prime septal (E/E) >15, ejection fraction < 50 percent (%), E deceleration time <= 150 millisecond (ms), isovolumic relaxation time (IVRT) <= 70 ms, any valve thickening (> trace regurgitation in mitral, aortic, pulmonary, or tricuspid valves), abnormal respiratory variation of inferior vena cava, pericardial effusion.
Time Frame: Baseline, Weeks 24, 48, and 72
Population: All participants who took at least 1 dose of tafamidis meglumine soft gelatin capsule 20 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis Meglumine 20 mg Once Daily (QD)
Number analyzed (Participants) | 15
Participants
  Number of Participants at Baseline | 9
  Number of Participants at Week 24 | 11
  Number of Participants at Week 48 | 9
  Number of Participants at Week 72 | 10

12. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: Protocol-required safety laboratory assessments include: Lymphocytes <0.8 × LLN; Neutrophils <0.8 × LLN, or >1.2 × ULN; Basophils >1.2 × ULN; Activated Partial Thromboplastin Time >1.1 × ULN; Prothrombin Time >1.1 × ULN; Prothrombin International Normalized Ratio >1.1 × ULN; Bilirubin >1.5 × ULN; Urate > 1.2 × ULN; Cholesterol >1.3 × ULN; Potassium <0.9 × LLN; Phosphate >1.2 × ULN; Bicarbonate >1.1 × ULN; Thyroid Stimulating Hormone >1.2 × ULN; URINE Protein ≥1; URINE Hemoglobin ≥1; Nitrite ≥1; URINE Erythrocytes ≥20; Epithelial Cells ≥6; and Casts >1.
Time Frame: Baseline up to Week 72
Population: All participants who took at least 1 dose of tafamidis meglumine soft gelatin capsule 20 mg
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis Meglumine 20 mg Once Daily (QD)
Number analyzed (Participants) | 15
Participants | 12

13. Secondary Outcome: Transthyretin (TTR) Concentrations on Day 1 (Baseline), and at Weeks 8, 12, 24, 48, and 72
Description: The TTR (also referred to as pre-albumin) concentrations were determined as pharmacodynamic (PD) biomarkers.
Time Frame: Baseline, Weeks 8, 12, 24, 48, and 72
Population: All participants who took at least 1 dose of tafamidis meglumine soft gelatin capsule 20 mg and who had at least 1 TTR concentration value.
Measure: Median (Full Range); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Tafamidis Meglumine 20 mg Once Daily (QD)
Number analyzed (Participants) | 15
Milligrams per deciliter (mg/dL)
  Median and Range of TTR Concentration on Day 1 (baseline) | 18.70 [9.03 to 28.0]
  Median and Range of TTR Concentration at Week 8: number analyzed (Participants) | 14
  Median and Range of TTR Concentration at Week 8 | 23.20 [13.5 to 36.2]
  Median and Range of TTR Concentration at Week 12 | 28.00 [13.5 to 33.3]
  Median and Range of TTR Concentration at Week 24 | 25.70 [13.3 to 30.9]
  Median and Range of TTR Concentration at Week 48: number analyzed (Participants) | 9
  Median and Range of TTR Concentration at Week 48 | 27.90 [19.0 to 33.4]
  Median and Range of TTR Concentration at Week 72: number analyzed (Participants) | 9
  Median and Range of TTR Concentration at Week 72 | 26.60 [14.4 to 32.2]

14. Secondary Outcome: TTR Stabilization and Percentage and 95% CI of Responders in TTR Stabilization at Post Baseline Visit
Description: The Fraction of Initial (FOI) is the ratio of the measured TTR tetramer concentration (post-denaturation) to the measured TTR concentration (pre-denaturation). Percent Stabilization (%) is the difference between the dosed FOI and the baseline FOI expressed as a percentage of the baseline FOI.
  Responder was the participant who achieved TTR stabilization (ie, who had been TTR stabilized). Percentage of responders was number of responders / number of evaluable (i.e., analyzed) participants.
Time Frame: Weeks 8, 12, 24, 48, and 72
Population: All participants who took at least 1 dose of tafamidis meglumine soft gelatin capsule 20 mg and who had at least 1 TTR stabilization value.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tafamidis Meglumine 20 mg Once Daily (QD)
Number analyzed (Participants) | 15
Percentage of participants
  Percentage and 95% CI of Responders in TTR Stabilization at Week 8: number analyzed (Participants) | 9
  Percentage and 95% CI of Responders in TTR Stabilization at Week 8 | 100.0 [66.4 to 100.0]
  Percentage and 95% CI of Responders in TTR Stabilization at Week 12: number analyzed (Participants) | 10
  Percentage and 95% CI of Responders in TTR Stabilization at Week 12 | 100.0 [69.2 to 100.0]
  Percentage and 95% CI of Responders in transthyretin (TTR) Stabilization at Week 24: number analyzed (Participants) | 10
  Percentage and 95% CI of Responders in transthyretin (TTR) Stabilization at Week 24 | 100.0 [69.2 to 100.0]
  Percentage and 95% CI of Responders in transthyretin (TTR) Stabilization at Week 48: number analyzed (Participants) | 6
  Percentage and 95% CI of Responders in transthyretin (TTR) Stabilization at Week 48 | 100.0 [54.1 to 100.0]
  Percentage and 95% CI of Responders in transthyretin (TTR) Stabilization at Week 72: number analyzed (Participants) | 8
  Percentage and 95% CI of Responders in transthyretin (TTR) Stabilization at Week 72 | 87.5 [47.3 to 99.7]

ADVERSE EVENTS:
Time Frame: Baseline up to Week 77
Arm/Group | Tafamidis Meglumine 20 mg Once Daily (QD)
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tafamidis Meglumine 20 mg Once Daily (QD) (N=15)
Amyloidosis (Immune system disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Orthostatic hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tafamidis Meglumine 20 mg Once Daily (QD) (N=15)
Anaemia (Blood and lymphatic system disorders) | 2
Coagulopathy (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Supraventricular extrasystoles (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Oedema peripheral (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
COVID-19 (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Compression fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 3
Ligament sprain (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Blood thyroid stimulating hormone decreased (Investigations) | 2
Electrocardiogram ST segment elevation (Investigations) | 1
Electrocardiogram abnormal (Investigations) | 1
Myoglobin blood increased (Investigations) | 1
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 1
Protein urine present (Investigations) | 1
QRS axis abnormal (Investigations) | 1
Total bile acids increased (Investigations) | 1
Urinary casts present (Investigations) | 1
Urinary occult blood positive (Investigations) | 1
Urinary sediment present (Investigations) | 2
White blood cell count decreased (Investigations) | 1
White blood cells urine positive (Investigations) | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hypozincaemia (Metabolism and nutrition disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Urethral haemorrhage (Renal and urinary disorders) | 1
Aortic arteriosclerosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT04828993/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT04828993/SAP_001.pdf